CLINICAL TRIAL: NCT03813394
Title: A Randomised Phase II Study of Pembrolizumab With or Without Bevacizumab in Platinum-resistant Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Bevacizumab and Pembrolizumab Combination in Platinum-resistant Recurrent/Metastatic NPC
Acronym: 2018/00947
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP01/2017/MSD3475
Record Dates: First submitted 2019-01-20; First posted 2019-01-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Locally Recurrent Cancer; Metastatic Nasopharyngeal Cancer
Keywords: Immunotherapy; Epstein Barr virus; Nasopharyngeal cancer; Anti-PD1; Tumor neoantigens
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections | interventions — pembrolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 into either Treatment Arm A or Arm B. Treatment will continue until tumor progression, intolerance to treatment, or up to 2 years (32 doses of pembrolizumab/bevacizumab). For patients who have progressed on pembrolizumab alone, cross over to Arm B is allowed, with repeat biopsy of the lesions before and 1 week after starting bevacizumab. Patients who discontinue from the trial will not be replaced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm A (Experimental): Intravenous pembrolizumab alone,D8 of 21-day cycle.
  Interventions: Drug: pembrolizumab
- Treatment Arm B (Experimental): Intravenous pembrolizumab preceded by an infusion of bevacizumab (Day 1 of 21-day cycle).
  Interventions: Drug: pembrolizumab; Drug: bevacizumab

INTERVENTIONS:
Drug: pembrolizumab — -Pembrolizumab in Solution for Injection
Drug: bevacizumab — * Bevacizumab in Concentrate for Solution
  * Bevacizumab in Concentrate for Solution
  Arms: Treatment Arm B

SUMMARY:
This is a single center, randomized, phase Ib/II open-label study of pembrolizumab (pembro or MK-3475) with or without bevacizumab in patients with recurrent non-curable or metastatic nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
The study will consist of 2 treatment arms. In Treatment Arm A, patients will be treated with intravenous pembrolizumab alone, 21-day cycle. For Treatment Arm B, patients will receive intravenous pembrolizumab preceded by an infusion of bevacizumab (Day 1 of 21-day cycle). Each treatment cycle is 3 weeks. Up to 48 patients will be enrolled in this study in 2 stages. The first stage will consist of 30 patients and the remaining 18 patients will be added if interim data looks promising.

Eligible patients will be randomized 1:1 into either Treatment Arm A or Arm B. Treatment will continue until tumor progression, intolerance to treatment, or up to 2 years (32 doses of pembrolizumab/bevacizumab). For patients who have progressed on pembrolizumab alone, cross over to Arm B is allowed, with repeat biopsy of the lesions before and 1 week after starting bevacizumab. Patients who discontinue from the trial will not be replaced.

The study will collect serial samples of tumor tissue and blood to determine the PD biomarkers of immune activation, in the tumor and systemically, following treatment. This is expected to provide preliminary evidence for immune stimulation using both pembrolizumab and bevacizumab in NPC. The tumor biopsies will also present an opportunity to determine the molecular details of tissue and tumor response to anti-angiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

- Participants are eligible to be included in the study only if all of the following criteria apply:

1. The participant (or legally acceptable representative if applicable) provides written consent for the trial.
2. Participants who are at least 21 years of age on the day of signing informed consent with histologically or cytologically confirmed diagnosis of non-keratinizing nasopharyngeal carcinoma (NPC) that has recurred at loco regional and/or distant sites will be enrolled in this study.
3. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Have locally or centrally determined EBV-positive NPC by EBV-encoded small RNA in situ hybridization (EBER in situ hybridization [ISH]) assay. If EBV-positive status has been previously determined by EBER ISH assay, then no re-testing is required. Note: If EBV status by EBER ISH assay has not been previously determined, tumor tissue from archival tissue may be submitted for EBV determination.
5. Received one or more lines of chemotherapy, which must include prior treatment with a platinum agent and must not be amenable to potentially curative radiotherapy or surgery.
6. Have provided archival tumor tissue sample of newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
7. Willingness to donate blood and tissue for mandatory translational research studies.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Have an adequate organ function.Specimens must be collected within 10 days prior to the start of study treatment.
10. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies: a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study medication.
11. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization. Note: Participants must have recovered from all AEs to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible. Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
2. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
3. Has a condition requiring systemic steroid therapy (> 10 mg daily prednisone equivalents) or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if < or = 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayedtype hypersensitivity reaction caused by contact allergen) is permitted.
4. Has a known history of active TB (Bacillus Tuberculosis).
5. Has had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, antiCTLA-4 antibody.
6. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
7. Has hypersensitivity to bevacizumab or any of its components.
8. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
9. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast or cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.
10. Has known brain metastases or leptomeningeal metastases, whether treated or untreated. NOTE: Primary nasopharyngeal cancers that directly invade the skull base and extend into the infratemporal fossa (e) are not regarded as brain metastases and are not excluded.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
18. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization/allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
19. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
20. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
21. Has received a live vaccine within 30 days of prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine.

Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint of ORR | 2 years
  Comparison of the two treatment arms will be evaluated using the Fisher's exact test. The treatment effect will be quantified via the relative risk estimate and its associated 95% confidence interval (CI).
The secondary endpoint of PFS | 2 years
  This will be summarized using the Kaplan-Meier survival estimate for each group. As an exploratory analysis, the log-rank test will be used for comparing differences in PFS, with its effect quantified based on hazard ratio and its 95% CI.
Progression free survival (PFS) | 2 years
  This is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded central imaging assessment or death due to any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be available, including data dictionaries, including all clinical data collected in the conduct of the trial in a deidentified format. Other documents available include the study protocol, statistical analysis plan, informed consent form and the clinical study report. This will be available beginning 3 months after article publication with no end date. Researchers whose proposed use of the data has been approved by an independent ethics review committee can access the data to achieve the aims in the proposal. Proposals should be directed to the corresponding author to provide data access following signing a data access agreement. The data will be made available by a link sent from the corresponding author to the requester.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: This will be available beginning 3 months after article publication with no end date.
Access Criteria: Researchers whose proposed use of the data has been approved by an independent ethics review committee can access the data to achieve the aims in the proposal. Proposals should be directed to the corresponding author to provide data access following signing a data access agreement. The data will be made available by a link sent from the corresponding author to the requester.

REFERENCES:
- [Background] Ma BB, Hui EP, Chan AT. Systemic approach to improving treatment outcome in nasopharyngeal carcinoma: current and future directions. Cancer Sci. 2008 Jul;99(7):1311-8. doi: 10.1111/j.1349-7006.2008.00836.x. Epub 2008 May 21. PMID 18498420
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Zarrabi K, Fang C, Wu S. New treatment options for metastatic renal cell carcinoma with prior anti-angiogenesis therapy. J Hematol Oncol. 2017 Feb 2;10(1):38. doi: 10.1186/s13045-016-0374-y. PMID 28153029
- [Derived] Chong WQ, Low JL, Tay JK, Le TBU, Goh GS, Sooi K, Teo HL, Cheo SW, Wong RT, Samol J, Lim MY, Li H, Shirgaonkar N, Chia S, Wang L, Gopinathan A, Eu DK, Tsang RK, Loh KS, Toh HC, Syn N, Kong LR, Dasgupta R, Tai BC, Lim YC, Goh BC. Pembrolizumab with or without bevacizumab in platinum-resistant recurrent or metastatic nasopharyngeal carcinoma: a randomised, open-label, phase 2 trial. Lancet Oncol. 2025 Feb;26(2):175-186. doi: 10.1016/S1470-2045(24)00677-6. Epub 2025 Jan 15. PMID 39826567